CLINICAL TRIAL: NCT05623865
Title: The Effect of Kinesio Taping on Edema Control and Wrist Functions in Conservatively Followed Distal Radius Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Levent Horoz, medical doctor, asisst prof, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAEK_
Record Dates: First submitted 2022-11-15; First posted 2022-11-21 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Distal Radius Fracture
Keywords: Distal Radius Fracture; kinesiotaping; edema
MeSH Terms: conditions — Wrist Fractures; Edema | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The person who evaluates the outcome criteria and the person who makes the interventions are different. The person who evaluates the outcome criteria is blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): After the initial evaluation, the patients will be randomly divided into two groups as the Experimental group and the control group.Experimental group will receive kinesiotape treatment in addition to those applied in the control group.
  Kinesiotape to the kinesio tape group will be done by a PM&R spesialist doctor who has a certificate of kinesiotaping, in accordance with the literature, using the lymphedema method.
  Interventions: Other: kinesiotaping; Other: exercise
- Control group (Other): Elevation and cold application, which is applied in the prevention and treatment of classical edema, will be recommended to the control group. In addition, wrist, elbow, finger range of motion and stretching exercises will be taught as a home exercise program.
  Interventions: Other: exercise

INTERVENTIONS:
Other: kinesiotaping — Kinesio tape will be attached with lymphedema technique.
  The bands will be removed prior to each assessment so that they do not affect the evaluator's blinding. After evaluation, the new tape will be fitted by the invesitgatör
  Arms: Experimental group
Other: exercise — Wrist, finger, elbow range of motion and stretching exercises will be taught to the patients and given as home exercises.
  In addition, patients will be given a leaflet containing illustrated and explanatory exercise visuals.

SUMMARY:
Kinesio tape is used successfully in the control of edema related to the extremity, especially in the control of lymphedema that develops after surgery.Kinesiotape is a non-allergic elastic tape applied to the skin surface.There are publications showing that kinesio tape applications are beneficial for edema control after interventional procedures such as anterior cruciate ligament surgery and knee prosthesis related to orthopedic surgical interventions. There is no publication on the effectiveness of kinesio tape application in the control and rehabilitation of post-cast edema of wrist fractures.It is planned to investigate the positive effects of kinesio tape in edema control and rehabilitation.

DETAILED DESCRIPTION:
The prevalence of distal radius fracture is increasing day by day. Circular cast is applied in 70-80% of patients treated for distal radius fractures.During the rehabilitation of patients after plaster application, joint stiffness, swelling on the hand and wrist, and edema are frequently encountered.Edema in the hand and wrist negatively affects the daily activities of patients, their quality of life, wrist and finger functions.

Edema is the main problem in rehabilitation after upper extremity injuries.It is known that fibrosis and adhesions in soft tissues develop as a result of prolonged extremity edema.

Elevation, massage, cold application, pressure gloves are used for edema control.

Kinesio tape is used successfully in the control of edema related to the extremity, especially in the control of lymphedema that develops after surgery.Kinesiotape is a non-allergic elastic tape applied to the skin surface. Kinesio Tape working mechanism opens the distance between the skin and subcutaneous tissues after it is applied to the skin and increases lymphatic drainage.

Kinesio tape also has the effect of supporting the joint and soft tissues around the joint.

Research on kinesio tape has generally focused on the control of lymphedema that develops after breast cancer surgery or stroke.

There are publications showing that kinesio tape applications are beneficial for edema control after interventional procedures such as anterior cruciate ligament surgery and knee prosthesis related to orthopedic surgical interventions.

Considering the studies conducted for edema control in patients treated for distal radius fractures, the effect of massage applications on edema has been investigated and it has been shown that massage has positive effects on edema control and wrist functions(9).

In another study, the effectiveness of modified massage methods in the treatment of edema was investigated and its positive effects were observed. There is no publication on the effectiveness of kinesio tape application in the control and rehabilitation of post-cast edema of wrist fractures. It is planned to investigate the positive effects of kinesio tape in edema control and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent plaster treatment for distal radius fracture
2. Patients over 18 years old

Exclusion Criteria:

1. To have been treated for lymphedema in the upper extremity before
2. Patients who have been operated for breast cancer
3. Bilateral distal raidus fracture
4. History of previous surgery related to the same extremity
5. Pathological fracture
6. Open fracture, active infection in the involved extremity
7. Presence of diseases with clinical course with peripheral edema such as heart failure, pulmonary hypertension
8. Cognitive dysfunction that impairs perception of test instructions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
volume measurement | 0 (baseline)
  The volume measurement of the patients after the cast will be measured with the upper extremity volumetric measuring device.
  The measurement will be made in comparison with each intact extremity. The measurement will be made standing up and at room temperature.Both extremity volume data will be recorded.
  The volume measurement of the patients after the cast will be measured with the upper extremity volumetric measuring device.The measurement will be made in comparison with each intact extremity. The measurement will be made standing up and at room temperature.
  Both extremity volume data will be recorded.
volume measurement | 5th day
  The volume measurement of the patients after the cast will be measured with the upper extremity volumetric measuring device.
  The measurement will be made in comparison with each intact extremity. The measurement will be made standing up and at room temperature.Both extremity volume data will be recorded.
  The volume measurement of the patients after the cast will be measured with the upper extremity volumetric measuring device.The measurement will be made in comparison with each intact extremity. The measurement will be made standing up and at room temperature.
  Both extremity volume data will be recorded.
volume measurement | 10th day
  The volume measurement of the patients after the cast will be measured with the upper extremity volumetric measuring device.
  The measurement will be made in comparison with each intact extremity. The measurement will be made standing up and at room temperature.Both extremity volume data will be recorded.
  The volume measurement of the patients after the cast will be measured with the upper extremity volumetric measuring device.The measurement will be made in comparison with each intact extremity. The measurement will be made standing up and at room temperature.
  Both extremity volume data will be recorded.
range of motion measurement | 0 (baseline)
  Wrist joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice.
  In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method.
range of motion measurement | 5th day
  Wrist joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice.
  In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method.
range of motion measurement | 10th day
  Wrist joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice.
  In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method.
Diameter Measurement | 0 (baseline)
  Both hands and wrists of the patient will be measured with the figure of eight method with the help of a tape measure.In addition, measurements will be made at the level of the bilateral wrist, metacarpophalangeal joint, and 6 cm proximal to the wrist.
Diameter Measurement | 5th day
  Both hands and wrists of the patient will be measured with the figure of eight method with the help of a tape measure.In addition, measurements will be made at the level of the bilateral wrist, metacarpophalangeal joint, and 6 cm proximal to the wrist.
Diameter Measurement | 10th day
  Both hands and wrists of the patient will be measured with the figure of eight method with the help of a tape measure.In addition, measurements will be made at the level of the bilateral wrist, metacarpophalangeal joint, and 6 cm proximal to the wrist.

SECONDARY OUTCOMES:
functionality | 0 (baseline)
  The short version of the Arm, Shoulder and Hand Questionnaire (Quick-DASH) Disability will be used to evaluate the functional status of the patients. Quick-DASH is a self-report questionnaire designed to measure physical function and symptoms in people with upper extremity musculoskeletal conditions. Turkish validity and reliability was established.
functionality | 5th day
  The short version of the Arm, Shoulder and Hand Questionnaire (Quick-DASH) Disability will be used to evaluate the functional status of the patients. Quick-DASH is a self-report questionnaire designed to measure physical function and symptoms in people with upper extremity musculoskeletal conditions. Turkish validity and reliability was established.
functionality | 10th day
  The short version of the Arm, Shoulder and Hand Questionnaire (Quick-DASH) Disability will be used to evaluate the functional status of the patients. Quick-DASH is a self-report questionnaire designed to measure physical function and symptoms in people with upper extremity musculoskeletal conditions. Turkish validity and reliability was established.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Horoz, Asisst Prof, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Ahi Evran University, Kirşehir, City Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crowe CS, Massenburg BB, Morrison SD, Chang J, Friedrich JB, Abady GG, Alahdab F, Alipour V, Arabloo J, Asaad M, Banach M, Bijani A, Borzi AM, Briko NI, Castle CD, Cho DY, Chung MT, Daryani A, Demoz GT, Dingels ZV, Do HT, Fischer F, Fox JT, Fukumoto T, Gebre AK, Gebremichael B, Haagsma JA, Haj-Mirzaian A, Handiso DW, Hay SI, Hoang CL, Irvani SSN, Jozwiak JJ, Kalhor R, Kasaeian A, Khader YS, Khalilov R, Khan EA, Khundkar R, Kisa S, Kisa A, Liu Z, Majdan M, Manafi N, Manafi A, Manda AL, Meretoja TJ, Miller TR, Mohammadian-Hafshejani A, Mohammadpourhodki R, Mohseni Bandpei MA, Mokdad AH, Naimzada MD, Ndwandwe DE, Nguyen CT, Nguyen HLT, Olagunju AT, Olagunju TO, Pham HQ, Pribadi DRA, Rabiee N, Ramezanzadeh K, Ranganathan K, Roberts NLS, Roever L, Safari S, Samy AM, Sanchez Riera L, Shahabi S, Smarandache CG, Sylte DO, Tesfay BE, Tran BX, Ullah I, Vahedi P, Vahedian-Azimi A, Vos T, Woldeyes DH, Wondmieneh AB, Zhang ZJ, James SL. Global trends of hand and wrist trauma: a systematic analysis of fracture and digit amputation using the Global Burden of Disease 2017 Study. Inj Prev. 2020 Oct;26(Supp 1):i115-i124. doi: 10.1136/injuryprev-2019-043495. Epub 2020 Mar 13. PMID 32169973
- [Background] Cheing GL, Wan JW, Kai Lo S. Ice and pulsed electromagnetic field to reduce pain and swelling after distal radius fractures. J Rehabil Med. 2005 Nov;37(6):372-7. doi: 10.1080/16501970510041055. PMID 16287669
- [Background] Knygsand-Roenhoej K, Maribo T. A randomized clinical controlled study comparing the effect of modified manual edema mobilization treatment with traditional edema technique in patients with a fracture of the distal radius. J Hand Ther. 2011 Jul-Sep;24(3):184-93; quiz 194. doi: 10.1016/j.jht.2010.10.009. Epub 2010 Dec 30. PMID 21193287
- [Background] Bell A, Muller M. Effects of kinesio tape to reduce hand edema in acute stroke. Top Stroke Rehabil. 2013 May-Jun;20(3):283-8. doi: 10.1310/tsr2003-283. PMID 23841976
- [Background] Tornatore L, De Luca ML, Ciccarello M, Benedetti MG. Effects of combining manual lymphatic drainage and Kinesiotaping on pain, edema, and range of motion in patients with total knee replacement: a randomized clinical trial. Int J Rehabil Res. 2020 Sep;43(3):240-246. doi: 10.1097/MRR.0000000000000417. PMID 32459670
- [Background] Haren K, Backman C, Wiberg M. Effect of manual lymph drainage as described by Vodder on oedema of the hand after fracture of the distal radius: a prospective clinical study. Scand J Plast Reconstr Surg Hand Surg. 2000 Dec;34(4):367-72. doi: 10.1080/028443100750059165. PMID 11195876